CLINICAL TRIAL: NCT07115550
Title: A Single-center, Single-arm, Phase II Clinical Study of Iparomlimab and Tuvonralimab Injection Combined With Regorafenib in the Treatment of Advanced Second-line or Above Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huai'an First People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY-2025-155-01
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Iparomlimab and Tuvonralimab; regorafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — regorafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iparomlimab and Tuvonralimab Injection combined with regorafenib (Experimental): Iparomlimab and Tuvonralimab Injection (QL1706): 5mg/kg,Q3W; Regorafenib:8mg(<60kg），12mg（≥60kg)
  Interventions: Drug: Iparomlimab and Tuvonralimab Injection (QL1706) in combination with Regorafenib

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab Injection (QL1706) in combination with Regorafenib — Iparomlimab and Tuvonralimab Injection (QL1706) in combination with Regorafenib

SUMMARY:
This study is a prospective, single-center, phase II clinical trial designed to evaluate the efficacy and safety of Iparomlimab and Tuvonralimab Injection (QL1706) combined with regorafenib in patients with advanced hepatocellular carcinoma (HCC) who have received at least one prior line of systemic therapy. The trial employs a single-arm design.

Study endpoint

Primary endpoint:

ORR

Secondary endpoint:

DCR, PFS, and OS evaluated based on RECIST v1.1. The incidence and severity of adverse events (AEs)

ELIGIBILITY:
Inclusion Criteria:

* 1. Volunteer to participate in this study and sign the informed consent form; 2. Age>=18 years old, male or female; 3. Unresectable advanced hepatocellular carcinoma confirmed by histopathology, cytology or imaging; 4. Have objective imaging progression during or after first-line treatment regimen or intolerance to first-line treatment regimen; 5. At least one measurable lesion according to the RESIST version 1.1 standard; 6. ECOG PS score: 0~1 points; 7. Child-Pugh liver function rating: A grade (<=6 points); 8. Expected survival time >=12 weeks; 9. Laboratory values within 3 days before the first dose meet the following requirements:

  1. Blood routine examination: (except for hemoglobin, no blood transfusion within 2 weeks prior to screening, no granulocyte colony-stimulating factor [G-CSF], no medication correction):

  <!-- -->

  1. Absolute neutrophil count >=1.5×10^9/L;
  2. Platelets >=75×10^9/L;
  3. Hemoglobin >=90 g/L; (2) Biochemical examination:

  <!-- -->

  1. Serum albumin >=30g/L;
  2. Serum total bilirubin <=1.5×ULN;
  3. ALT and AST <=3×ULN;
  4. Serum creatinine <=1.5×ULN; or Cr clearance > 50 mL/min (3) International normalized ratio (INR) <=1.2 or prothrombin time (PT) above the range of normal controls <=2 seconds; (4) Urine protein <2 (if urine protein >=2, 24-hour (h) urine protein quantification can be performed, and 24-hour urine protein quantification <1.0g can be enrolled); 10. If you have hepatitis B virus (HBV) infection, such as HBsAg positive, HBV-DNA needs to be tested, and HBV-DNA needs to be < 2000 IU/mL (if the study center only has copy/mL testing units, it must be <104 copy/mL); For subjects with HBV-DNA>=2000 IU/mL, receive at least 1 week of antiviral therapy (only nucleosides such as entecarvir, tenofovir fumarate, and propofol tenofovir fumarate tablets) are allowed, and viral copy number decreases by more than 10 times (1 lg) compared to before the first dose. For HBV-infected patients, antiviral therapy is required throughout the study. Hepatitis C virus (HCV)-RNA-positive subjects must receive antiviral therapy as per treatment guidelines; 11. Women of childbearing age must have a negative pregnancy test (βHCG) before starting the first dose. Women of childbearing potential and men (who have sex with women of childbearing potential) must agree to use contraception during treatment and for 6 months of the last dose.

Exclusion Criteria:

* 1. Known cases of fibroblastic layer HCC, sarcomatoid HCC or mixed-type cholangiocarcinoma and HCC; 2. Prior to the first dose of the study treatment, there was toxicity that did not recover to the 5.0 version of the National Cancer Institute Common Toxicity Criteria (NCI CTCAEv5.0) level 1 (excluding hair loss, non-clinically significant and asymptomatic laboratory abnormalities); 3. History of hepatic encephalopathy, hepatorenal syndrome or more severe liver cirrhosis of Child-Pugh B grade; 4. Imaging shows portal vein invasion of the main portal branch (Vp4), inferior vena cava or hepatocellular carcinoma involving the heart; 5. Previously received regorafenib treatment; 6. Within 5 years before the first administration, there was a history of malignant tumor other than HCC, with a negligible risk of metastasis or death (such as 5-year OS rate > 90%), such as well-treated cervical carcinoma in situ, non-melanoma skin cancer, localized prostate cancer, ductal carcinoma in situ, or stage I uterine cancer; 7. Coinfection with HBV and HCV, or co-infection with HBV and delta hepatitis virus; 8. History of idiopathic pulmonary fibrosis, organizing pneumonia (such as obliterative bronchiolitis), drug-induced pneumonia or idiopathic pneumonia, or screening chest CT scan shows evidence of active pneumonia; 9. Active tuberculosis; 10. History of autoimmune diseases or immunodeficiency diseases, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener's granulomatosis, Sjogren's syndrome, Guillain-Barré syndrome or multiple sclerosis; 11. Within 4 weeks before the first administration, had a severe infection, including but not limited to hospitalization due to infection complications, bacteremia or severe pneumonia; 12. Received oral or intravenous antibiotic therapy within 2 weeks before the first dose; 13. Use of nonsteroidal anti-inflammatory drugs (NSAIDs) for daily treatment of chronic diseases; 14. Evidence of bleeding diathesis or significant coagulation dysfunction (not receiving anticoagulant therapy); 15. Current or recent use of aspirin or full-dose oral or intravenous anticoagulants; 16. Bleeding events due to untreated or incompletely treated esophageal and/or gastric varices within 6 months prior to the first dose; 17. Major vascular disease (such as aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months before the first dose; 18. Inadequately controlled arterial hypertension (systolic blood pressure>=140mmHg or diastolic blood pressure >=90mmHg) (based on the average of BP readings obtained from >=2 measurements), allowing the above parameters to be achieved by antihypertensive therapy; Previous hypertensive crisis or hypertensive encephalopathy; 19. Significant uncontrolled or symptomatic hypercalcemia (ionized calcium >1.5mmol/L, calcium >12 mg/dL, or corrected serum calcium >ULN) before the first dose; 20. Severe cardiovascular disease (such as New York Heart Association Class II or above, myocardial infarction, or cerebrovascular accident), unstable arrhythmia, or unstable angina within 3 months; 21. Clinically significant ascites; 22. History of intra-abdominal inflammation in the 6 months prior to the first dose, including but not limited to peptic ulcer, diverticulitis, or colitis; 23. History of abdominal or tracheoesophageal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months before the first dose; 24. Severe, non-healing or dehisced wound, active ulcer, or untreated bone fracture; 25. Hollow needle biopsy or other minor surgery within 3 days prior to the first dose, excluding placement of vascular access devices; 26. Major surgery within 4 weeks prior to the first dose of medication, or anticipation of need for major surgery during the study; 27. Treatment with systemic immunosuppressive drugs (including but not limited to glucocorticoids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor-α [TNF-α preparations) within 2 weeks prior to the first dose, or those who are expected to need systemic immunosuppressive drugs during the study treatment; 28. Subjects who have received or will receive a live vaccine within 30 days before the first dose, or who need to use the vaccine during the expected treatment period or within 5 months after the last dose; 29. Known allergy to any of the study drugs or excipients; 30. Women who are contraindicated to use an investigational drug, any other disease that may affect the interpretation of the results or may place the patient at high risk of treatment complications, metabolic dysfunction, physical examination findings, or clinical laboratory findings that are pregnant, lactating, have given birth but refuse to use contraception; 31. Other factors that the investigator deems unsuitable for participation in the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-08-26 (Estimated); Primary Completion 2027-08-26 (Estimated); Study Completion 2028-08-26 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | At the end of Cycle 6 (each cycle is 21 days)